CLINICAL TRIAL: NCT06596486
Title: A Comparison of CoolStick and Ethyl Chloride Spray for the Assessment of Sensory Block to Light Touch and Cold Before Caesarean Section Under Spinal or Combined Spinal-epidural Anaesthesia
Brief Title: A Comparison of CoolStick With Ethyl Chloride for the Assessment of Light Touch
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 331686
Record Dates: First submitted 2024-08-22; First posted 2024-09-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ethyl Chloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All participants will receive standard care with the addition of extra assessment of block from neuraxial anaesthesia
  Interventions: Other: CoolStick; Other: Ethyl Chloride; Other: Question

INTERVENTIONS:
Other: CoolStick — Assessment of block using CoolStick.
Other: Ethyl Chloride — Assessment of block using ethyl chloride spray
Other: Question — Participant will be asked if they felt pain or not.

SUMMARY:
The main aim of this study is to compare CoolStick to ethyl chloride spray for the assessment of light touch following neuraxial anaesthesia for caesarean delivery.

Coolstick and ethyl chloride will also be compared for the assessment of cold sensation.

Participants will also be asked whether they experienced any intraoperative pain.

DETAILED DESCRIPTION:
In England, up to 35% of deliveries in 2022 were by caesarean section. Current guidelines from NICE recommend that regional anaesthesia is offered for caesarean section. Neuraxial anaesthesia is considered to carry less risk of morbidity than general anaesthesia for both mother and neonate and is performed for approximately 92% of caesarean sections. To ensure the comfort of the mother, and to avoid intraoperative pain that could lead to general anaesthesia conversion, the neuraxial block is tested prior to commencing surgery. In the United Kingdom, the Royal College of Anaesthetists recommend that less than 1% of elective caesarean sections started under regional anaesthesia are converted to general anaesthesia.

Surveys of UK anaesthetists have found a wide range of practices when assessing neuraxial block, including the testing of light touch, temperature, pain and motor block. In a survey of UK anaesthetists, cold has been shown to be the most widely used modality for testing with 92% of respondents testing this modality. This was followed by touch, which 60% of respondents tested for. Recent consensus guidance from the Obstetric Anaesthetists' Association has recommended light touch as the primary testing modality for neuraxial anaesthesia for caesarean section, aiming for a sensory block to the T5 level or above. A second testing modality is recommended in cases where there is doubt over the light touch assessment. In practice, many anaesthetists will consider anaesthesia to be adequate when block to light touch is demonstrated to the T5 level or above and cold to the T4 level or above.

Ethyl chloride spray is the most common piece of equipment for used for testing in the UK. It has been shown that ethyl chloride spray can be used for the assessment of light touch and is equivalent to established methods when assessing adequacy of the block for surgery. However, ethyl chloride has disadvantages: skin irritation and allergic reactions sometimes occur; and containers are expensive, require replacing and carry a carbon footprint. The spray also remains in the atmosphere for up to two months and this can have a deleterious effect on the environment.

Cotton wool has been shown to be as effective at testing light touch when compared to more expensive methods. However, it is not necessarily practical to have multiple pieces of equipment required to assess different block modalities. Given that ethyl chloride is commonly used to test both modalities, a more sustainable and cost-effective approach to testing both light touch and cold would be ideal.

Theophany Limited recently developed the CoolStick for assessment of block height to cold. The CoolStick consists of a stainless-steel head and a plastic handle. It is kept in the fridge before use and is cleaned with an antibacterial wipe between patients. The CoolStick maintains a temperature adequate for cold assessment for up to 10 minutes in ambient theatre temperature and should be kept refrigerated for at least 40 minutes prior to use. It appears to be a more sustainable and cost-effective alternative to ethyl chloride spray; however, there are no studies that demonstrate its clinical application in this setting.

The primary aim of this study is to compare Coolstick with ethyl chloride spray for the assessment of light touch, with the secondary aim of comparing CoolStick to ethyl chloride for the assessment of cold.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients presenting for elective caesarean section under spinal or combined spinal-epidural anaesthesia.

Exclusion Criteria:

* < 18 years old
* Unwilling or unable to give informed consent
* Inability to understand written and/or verbal English
* Allergy to stainless steel
* Allergy to ethyl chloride spray

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All eligible patients presenting for elective caesarean section will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Light Touch | 6 months
  The dermatomal block level to light touch at 10 minutes after spinal injection measured using CoolStick and Ethyl Chloride spray.

SECONDARY OUTCOMES:
Cold | 6 months
  The dermatomal block level to cold at 10 minutes after spinal injection measured using CoolStick and Ethyl Chloride spray.

OTHER OUTCOMES:
Intraoperative pain | 6 months
  The presence of intraoperative pain within 60 minutes of the spinal injection. The options will be 'yes' or 'no'.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wikner, Study Chair — Barts & The London NHS Trust
Locations (3):
- United Kingdom (3):
  - Newham University Hospital, London
  - The Royal London Hospital, London
  - Whipps Cross University Hospital, London

IPD SHARING:
Plan to Share IPD: No